CLINICAL TRIAL: NCT03986580
Title: Prospective Evaluation Of Lumbar Discectomy With Additional Implantation Of An Annular Closure Device In Patients With Large Postsurgical Annular Defects For Prevention Of Lumbar Disc Reherniation
Brief Title: Study of Lumbar Discectomy With Annular Closure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Intrinsic Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-010
Record Dates: First submitted 2019-06-06; First posted 2019-06-14 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Annular closure device (Other): Single arm study; all patients treated with an annular closure device
  Interventions: Device: Annular closure device

INTERVENTIONS:
Device: Annular closure device — Annular closure, following limited discectomy procedure at a single LS level between L4 and S1

SUMMARY:
The purpose of this prospective, single-arm, multicenter study is to assess an annular closure device when used as an adjunct to a primary lumbar limited discectomy, to limited discectomy alone.

DETAILED DESCRIPTION:
This single-arm case series will enroll 75 patients at select US (approximately 8-10) sites. Patients that are scheduled for a single-level L4-S1 discectomy and who meet the pre-operative eligibility criteria will be considered for study participation. Patients that meet all intraoperative criteria will be enrolled into the study and treated with lumbar discectomy and additional annular closure device implantation. All enrolled subjects will be followed for at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old and skeletally mature (male or female)
2. Subjects with posterior or posterolateral disc herniations at one level between L4 and S1 with radiographic confirmation of neural compression using MRI. [Note: Intraoperatively, only patients with an anular defect (post discectomy) between 4mm and 6mm tall and 6mm and 10mm wide shall qualify.]
3. At least six (6) weeks of failed, conservative treatment prior to surgery, including physical therapy, use of anti-inflammatory medications at maximum specified dosage and/or administration of epidural/facet injections.;
4. Minimum posterior disc height of 5mm at the index level.
5. Radiculopathy (with or without back pain) with a positive Straight Leg Raise (0 - 60 degrees)
6. Oswestry Questionnaire score of at least 40/100 at baseline.
7. VAS leg pain (one or both legs) of at least 40/100 at baseline.
8. Psychosocially, mentally and physically able to fully comply with the clinical protocol and willing to adhere to follow-up schedule and requirements.

Exclusion Criteria:

1. Spondylolisthesis Grade II or higher (25% slip or greater).
2. Subject requires spinal surgery other than a discectomy (with or without laminotomy) to treat leg/back pain (scar tissue and osteophyte removal is allowed).
3. Subject has back or non-radicular leg pain of unknown etiology.
4. Prior surgery at the index lumbar vertebral level
5. Subject requiring a spine DEXA (i.e., patients with SCORE of ≥ 6) with a T Score less than -2.0 at the index level. For patients with a herniation at L5/S1, the average T score of L1-L4 shall be used.
6. Subject has clinically compromised vertebral bodies in the lumbosacral region due to any traumatic, neoplastic, metabolic, or infectious pathology.
7. Subject has sustained pathologic fractures of the vertebra or multiple fractures of the vertebra or hip
8. Subject has scoliosis of greater than ten (10) degrees (both angular and rotational).
9. Any metabolic bone disease.
10. Subject has an active infection either systemic or local.
11. Subject has cauda equina syndrome or neurogenic bowel/bladder dysfunction.
12. Subject has severe arterial insufficiency of the legs or other peripheral vascular disease. (Screening on physical examination for patients with diminution or absence of dorsalis pedis or posterior tibialis pulses. If diminished or absent by palpation, then an arterial ultrasound is required with vascular plethysmography. If the absolute arterial pressure is below 50mm of Hg at the calf or ankle level, then the patient is to be excluded.)
13. Subject has significant peripheral neuropathy, defined as a subject with Type I or Type II diabetes or similar systemic metabolic condition causing decreased sensation in a stocking-like or non-radicular and non-dermatomal distribution in the lower extremities.
14. Subject has insulin-dependent diabetes mellitus.
15. Subject is morbidly obese (defined as a body mass index >40, or weighs more than 100 lbs over ideal body weight).
16. Subject has been diagnosed with active hepatitis, AIDS, or HIV.
17. Subject has been diagnosed with rheumatoid arthritis or other autoimmune disease.
18. Subject has a known allergy to titanium, polyethylene or polyester materials.
19. Any subject that cannot have a baseline MRI taken.
20. Subject is pregnant or interested in becoming pregnant in the next 2 years.
21. Subject has active tuberculosis or has had tuberculosis in the past three (3) years.
22. Subject has a history of active malignancy: A subject with a history of any invasive malignancy (except non-melanoma skin cancer), unless he/she has been treated with curative intent and there have been no signs or symptoms of the malignancy for at least two (2) years.
23. Subject is immunologically suppressed, received steroids >1 month over the past year.
24. Currently taking anticoagulants, other than aspirin, unless the patient can be taken off the anticoagulant for surgery.
25. Subject has a current chemical/alcohol dependency or significant psychosocial disturbance.
26. Subject has a life expectancy of less than three (3) years.
27. Subject is currently involved in active spinal litigation.
28. Subject is currently involved in another investigational study.
29. Subject is incarcerated.
30. Any contraindication for MRI (e.g. claustrophobia, contrast allergy).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Blood loss | Intra-operative
  Amount of blood loss measured in ml
Procedure time | Intra-operative
  Length of surgery, measured in minutes
Hospital stay | Post-procedure hospital discharge day (in average between 1 and 3 days post surgery)
  Length of the hospital stay measured in days between hospital admission and hospital discharge
Discharge status | Post-procedure hospital discharge day (in average between 1 and 3 days post surgery)
  Evaluation of improvement in motor and sensory neurologic status
Leg pain severity (0-100 VAS score) | Baseline, 4 Weeks, 3 Months, 1 year
  Change from baseline of Visual Analogue Scale score (values between 0-100), with lower values representing better outcome
Back pain severity (0-100 VAS score) | Baseline, 4 Weeks, 3 Months, 1 year
  Change from baseline of Visual Analogue Scale score (values between 0-100), with lower values representing better outcome
ODI | Baseline, 4 Weeks, 3 Months, 1 year
  Change from baseline in Oswestry Disability Index. The ODI is scored on a scale from 0% to 100%, with higher scores indicating higher levels of disability
EQ-5D | Baseline, 4 Weeks, 3 Months, 1 year
  Change from baseline in EQ-5D. The EuroQol (EQ-5D) is a generic utility measure used to characterize current health states. The subject-reported questionnaire consists of 5 domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each of which can take one of three responses. Possible responses include three levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D dimension
Satisfaction with surgery procedure | 1 year
  Patient satisfaction with surgery and treatment assessed utilizing questionnaire with Composite questionnaire with 2 questions will be administered; 1.) Indicate degree of satisfaction with the outcome and 2.) likelihood of recommending the procedure to others
Neurological assessment | Baseline, 4 Weeks, 3 Months, 1 year
  Change from baseline in sensory (sensation response at dermatomal levels) reflex, (knee jerk, ankle jerk, response measured as "normal", "increased", "absent" and "decreased") and muscle strength measured 0-5 with "0" representing no evidence of motor strength and "5" representing full resistance
Adverse events | Baseline, Intra-operative, 4 Weeks, 3 Months, 1 year
  Change of health status with occurrence of adverse event, reported by seriousness and relationship to the device or procedure
Hospital readmission occurrence | Post-procedure hospital discharge day (in average between 1 and 3 days post surgery), 4 Weeks, 3 Months, 1 year
  Change from baseline in incidence of re-admissions to hospital, post treatment
Symptomatic reherniation incidence | Post-procedure hospital discharge day (in average between 1 and 3 days post surgery), 4 Weeks, 3 Months, 1 year
  Change from baseline in incidence of post-operative recurrent herniation at the index level. Recurrent herniation may be confirmed surgically, or radiographically as determined by an independent review
Reoperation incidence | Post-procedure hospital discharge day (in average between 1 and 3 days post surgery), 4 Weeks, 3 Months, 1 year
  Change from baseline in incidence of post-operative reoperation at the index level
Return to work assessment | 4 Weeks, 3 Months, 1 year
  Change from baseline in work status (ability to return to work, with or without reported restrictions)
Opioid consumption | Baseline, Intra-operative, Post-procedure hospital discharge day (in average between 1 and 3 days post surgery), 4 Weeks, 3 Months, 1 year
  Change from baseline for all opioid based medications (routes of administration (oral, IV, transdermal), dosing (mg/ml/tablet), duration (days)).

CONTACTS AND LOCATIONS:
Overall Officials: David H Kim, MD, Study Chair — New England Baptist Hospital
Locations (7):
- United States (7):
  - UC San Diego Health System, San Diego, California
  - Baptist - Lyerly Neurosurgery, Jacksonville, Florida
  - North Shore University Health System, Evanston, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - Louisiana Spine Institute, Shreveport, Louisiana
  - Salt Lake Orthopaedic Clinic, Salt Lake City, Utah

REFERENCES:
- [Derived] Strenge KB, DiPaola CP, Miller LE, Hill CP, Whitmore RG. Multicenter study of lumbar discectomy with Barricaid annular closure device for prevention of lumbar disc reherniation in US patients: A historically controlled post-market study protocol. Medicine (Baltimore). 2019 Aug;98(35):e16953. doi: 10.1097/MD.0000000000016953. PMID 31464935